CLINICAL TRIAL: NCT04612881
Title: Clinical Verification of the Activity and Tolerability of Fitostimoline Vaginal Pessaries in Women With Hysterectomy. Randomized, Perspective, Monoscentric Study.
Brief Title: Fitostimoline Vaginal Pessaries in Women With Hysterectomy. Randomized, Perspective, Monoscentric Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Vignali, PROFESSOR, University of Milan
Other Study IDs: Fitostimoline pessaries
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Vaginal Bleeding
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- fitostimoline vaginal pessaries
  Interventions: Drug: fitostimoline vaginal pessaries; Other: standard of care

INTERVENTIONS:
Drug: fitostimoline vaginal pessaries — vaginal pessaries
Other: standard of care — standard of care

SUMMARY:
Clinical evaluation of Fitostimoline vaginal pessaries in the treatment of hysterectomy. An observational, randomized, perspective study performed on 60 women where 30 women are treated with fitostimoline pessaries and 30 women are treated with the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patient aged between 35 and 80 years
* patient undergoing hysterectomy
* Willingness to understand the procedures and aims of the study

Exclusion Criteria:

* Anamnestic or clinical data of metabolic or endocrine diseases (such as uncontrolled diabetes mellitus) or any other local and / or systemic pathology potentially able to interfere with the study parameters;
* Concomitant treatment with antibiotics / antiseptics, NSAIDs, analgesics (excl. Paracetamol)
* Non-therapeutic use of psychoactive substances;
* Abuse of drugs and / or alcohol / smoking;
* Neurological disorders or psychiatric conditions potentially capable of affecting the validity of the consent and / or compromising the patient's adherence to the study procedures;
* Known allergy, hypersensitivity or intolerance to the constituents of the preparations under study;
* Any condition, medical or otherwise, that could significantly reduce the possibility of obtaining reliable data, achieving the objectives of the study, perfecting its completion;
* Presumption of poor reliability or collaboration;
* Treatment with any preparation in the last 30 days prior to the start of the study;
* Patients already enrolled in this study;
* Center staff directly involved in the study and close relatives

Ages: 30 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Study Population: women aged between 30 and 80 years with hysterctomy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-18 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2021-09-18 (Estimated)

PRIMARY OUTCOMES:
TSS | 60 days
  total symptom score (TSS) on a scale from 0 to 10 from worst to best

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Maglione, Napoli, Italy